CLINICAL TRIAL: NCT01263197
Title: Effect of LY2216684 on Heart Rate and Blood Pressure in Healthy Subjects Receiving Oral Doses of Albuterol or Propranolol
Brief Title: A Study of LY2216684 in Healthy Participants Receiving Albuterol or Propanolol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12598; H9P-EW-LNCI (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Albuterol; Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY2216684, albuterol, LY2216684+albuterol (Experimental): LY2216684 as an 18 milligram (mg) oral dose on days 1-5 and placebo for albuterol on days 1, 3 and 5 in first intervention period, placebo for LY2216684 on days 1-5 and albuterol as a 2 mg oral dose on days 1, 3 and 5 in the second intervention period, and LY2216684 as an 18 mg oral dose on days 1-5 and albuterol as a 2 mg oral dose on days 1, 3 and 5 in the third intervention period. There is a minimum 7 day washout between each intervention period.
  Interventions: Drug: LY2216684; Drug: albuterol; Drug: placebo for LY2216684; Drug: placebo for albuterol
- albuterol, LY2216684+albuterol, LY2216684 (Experimental): Placebo for LY2216684 on days 1-5 and albuterol as a 2 mg oral dose on days 1, 3 and 5 in the first intervention period, LY2216684 as an 18 mg oral dose on days 1-5 and albuterol as a 2 mg oral dose on days 1, 3 and 5 in the second intervention period, and LY2216684 as an 18 mg oral dose on days 1-5 and placebo for albuterol on days 1, 3 and 5 in third intervention period. There is a minimum 7 day washout between each intervention period.
  Interventions: Drug: LY2216684; Drug: albuterol; Drug: placebo for LY2216684; Drug: placebo for albuterol
- LY2216684+albuterol, LY2216684, albuterol (Experimental): LY2216684 as an 18 mg oral dose on days 1-5 and albuterol as a 2 mg oral dose on days 1, 3 and 5 in the first intervention period, LY2216684 as an 18 mg oral dose on days 1-5 and placebo for albuterol on days 1, 3 and 5 in second intervention period, Placebo for LY2216684 on days 1-5 and albuterol as a 2 mg oral dose on days 1, 3 and 5 in the third intervention period. There is a minimum 7 day washout between each intervention period.
  Interventions: Drug: LY2216684; Drug: albuterol; Drug: placebo for LY2216684; Drug: placebo for albuterol
- LY2216684, propranolol, LY2216684+propranolol (Experimental): LY2216684 as an 18 mg oral dose on days 1-5 and placebo for propranolol on days 1, 3 and 5 in first intervention period, placebo for LY2216684 on days 1-5 and propranolol as a 40 mg oral dose on days 1, 3 and 5 in the second intervention period, and LY2216684 as an 18 mg oral dose on days 1-5 and propranolol as a 40 mg oral dose on days 1, 3 and 5 in the third intervention period. There is a minimum 7 day washout between each intervention period.
  Interventions: Drug: LY2216684; Drug: propranolol; Drug: placebo for LY2216684; Drug: placebo for propranolol
- propranolol, LY2216684+propranolol, LY2216684 (Experimental): Placebo for LY2216684 on days 1-5 and propranolol as a 40 mg oral dose on days 1, 3 and 5 in the first intervention period, LY2216684 as an 18 mg oral dose on days 1-5 and propranolol as a 40 mg oral dose on days 1, 3 and 5 in the second intervention period, and LY2216684 as an 18 mg oral dose on days 1-5 and placebo for propranolol on days 1, 3 and 5 in third intervention period. There is a minimum 7 day washout between each intervention period.
  Interventions: Drug: LY2216684; Drug: propranolol; Drug: placebo for LY2216684; Drug: placebo for propranolol
- LY2216684+propranolol, LY2216684, propranolol (Experimental): LY2216684 as an 18 mg oral dose on days 1-5 and propranolol as a 40 mg oral dose on days 1, 3 and 5 in the first intervention period, LY2216684 as an 18 mg oral dose on days 1-5 and placebo for propranolol on days 1, 3 and 5 in second intervention period, placebo for LY2216684 on days 1-5 and propranolol as a 40 mg oral dose on days 1, 3 and 5 in the third intervention period. There is a minimum 7 day washout between each intervention period.
  Interventions: Drug: LY2216684; Drug: propranolol; Drug: placebo for LY2216684; Drug: placebo for propranolol

INTERVENTIONS:
Drug: LY2216684 — administered orally
Drug: albuterol — administered orally
  Arms: LY2216684+albuterol, LY2216684, albuterol; LY2216684, albuterol, LY2216684+albuterol; albuterol, LY2216684+albuterol, LY2216684
Drug: propranolol — administered orally
  Arms: LY2216684+propranolol, LY2216684, propranolol; LY2216684, propranolol, LY2216684+propranolol; propranolol, LY2216684+propranolol, LY2216684
Drug: placebo for LY2216684 — administered orally
Drug: placebo for albuterol — administered orally
  Arms: LY2216684+albuterol, LY2216684, albuterol; LY2216684, albuterol, LY2216684+albuterol; albuterol, LY2216684+albuterol, LY2216684
Drug: placebo for propranolol — administered orally
  Arms: LY2216684+propranolol, LY2216684, propranolol; LY2216684, propranolol, LY2216684+propranolol; propranolol, LY2216684+propranolol, LY2216684

SUMMARY:
The purpose of this study is to determine the effect of LY2216684 on heart rate of participants receiving Albuterol and Propranolol. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy, as determined by medical history and physical examination.
* Male participants - Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.
* Female participants - Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or Women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause [at least 1 year without menses or 6 months without menses and a follicle stimulating hormone (FSH) >40 milli-international units per milliliter (mIU/mL)].
* Have a body weight >50 kilograms (kg).
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Have normal blood pressure and pulse rate (sitting position) as determined by the investigator.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device other than the study drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2216684, albuterol (Group 1 only), propranolol (Group 2 only), or related compounds.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to screening.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have a history of or current asthma, including exercise induced asthma.
* Have a history or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Intend to use over-the-counter or prescription medication (including hormonal contraceptives) within 14 days prior to dosing unless deemed acceptable by the investigator and Sponsor's medical monitor
* Have donated blood of more than 500 milliliters (mL) within the last month.
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption 48 hours prior to check-in in each period and while resident at the Clinical Research Unit (CRU) [1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits].
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participants unwilling to adhere to study caffeine restrictions.
* Have used any tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment and during the study.
* Have a documented or suspected history of glaucoma.
* Participants determined to be unsuitable by the investigator for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 3-period, crossover study conducted in 2 groups. Participants were randomized to 1 of 3 sequences in either the albuterol group (Group 1) or 1 of 3 sequences in the propranolol group (Group 2).
Groups:
- Group 1, Seq 1: LY2216684, Albuterol, LY2216684+Albuterol: Group 1, Sequence (Seq) 1
  First intervention: LY2216684 administered as an 18-milligram (mg) oral dose (two 9-mg tablets) once daily (QD) on Days 1 through 5 with single oral doses of placebo (for albuterol) co-administered on Days 1, 3, and 5.
  Second intervention: Oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5.
  Third intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5.
  There was a minimum 7-day washout between each intervention period.
- Group 1, Seq 2: Albuterol, LY2216684+Albuterol, LY2216684: Group 1, Sequence 2
  First intervention: Oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5.
  Second intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5.
  Third intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of placebo (for albuterol) co-administered on Days 1, 3, and 5.
  There was a minimum 7-day washout between each intervention period.
- Group 1, Seq 3: LY2216684+Albuterol, LY2216684, Albuterol: Group 1, Sequence 3
  First intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5.
  Second intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of placebo (for albuterol) co-administered on Days 1, 3, and 5.
  Third intervention: Oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5.
  There was a minimum 7-day washout between each intervention period.
- Group 2, Seq 1: LY2216684, Propranolol, LY2216684+Propranolol: Group 2, Sequence 1
  First intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of placebo (for propranolol) co-administered on Days 1, 3, and 5.
  Second intervention: Oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 40 mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5.
  Third intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of 40 mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5.
  There was a minimum 7-day washout between each intervention period.
- Group 2, Seq 2: Propranolol, LY2216684+Propranolol, LY2216684: Group 2, Sequence 2
  First intervention: Oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 40 mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5.
  Second intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of 40 mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5.
  Third intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of placebo (for propranolol) co-administered on Days 1, 3, and 5.
  There was a minimum 7-day washout between each intervention period.
- Group 2, Seq 3: LY2216684+Propranolol, LY2216684, Propranolol: Group 2, Sequence 3
  First intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of 40 mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5.
  Second intervention: LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of placebo (for propranolol) co-administered on Days 1, 3, and 5.
  Third intervention: Oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 40 mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5.
  There was a minimum 7-day washout between each intervention period.
Period: First Intervention (Period 1)
Arm/Group | Group 1, Seq 1: LY2216684, Albuterol, LY2216684+Albuterol | Group 1, Seq 2: Albuterol, LY2216684+Albuterol, LY2216684 | Group 1, Seq 3: LY2216684+Albuterol, LY2216684, Albuterol | Group 2, Seq 1: LY2216684, Propranolol, LY2216684+Propranolol | Group 2, Seq 2: Propranolol, LY2216684+Propranolol, LY2216684 | Group 2, Seq 3: LY2216684+Propranolol, LY2216684, Propranolol
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout Period 1
Arm/Group | Group 1, Seq 1: LY2216684, Albuterol, LY2216684+Albuterol | Group 1, Seq 2: Albuterol, LY2216684+Albuterol, LY2216684 | Group 1, Seq 3: LY2216684+Albuterol, LY2216684, Albuterol | Group 2, Seq 1: LY2216684, Propranolol, LY2216684+Propranolol | Group 2, Seq 2: Propranolol, LY2216684+Propranolol, LY2216684 | Group 2, Seq 3: LY2216684+Propranolol, LY2216684, Propranolol
Started | 8 | 8 | 8 | 8 | 8 | 7
Completed | 8 | 8 | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Period: Second Intervention (Period 2)
Arm/Group | Group 1, Seq 1: LY2216684, Albuterol, LY2216684+Albuterol | Group 1, Seq 2: Albuterol, LY2216684+Albuterol, LY2216684 | Group 1, Seq 3: LY2216684+Albuterol, LY2216684, Albuterol | Group 2, Seq 1: LY2216684, Propranolol, LY2216684+Propranolol | Group 2, Seq 2: Propranolol, LY2216684+Propranolol, LY2216684 | Group 2, Seq 3: LY2216684+Propranolol, LY2216684, Propranolol
Started | 8 | 8 | 8 | 8 | 7 | 7
Completed | 8 | 8 | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Group 1, Seq 1: LY2216684, Albuterol, LY2216684+Albuterol | Group 1, Seq 2: Albuterol, LY2216684+Albuterol, LY2216684 | Group 1, Seq 3: LY2216684+Albuterol, LY2216684, Albuterol | Group 2, Seq 1: LY2216684, Propranolol, LY2216684+Propranolol | Group 2, Seq 2: Propranolol, LY2216684+Propranolol, LY2216684 | Group 2, Seq 3: LY2216684+Propranolol, LY2216684, Propranolol
Started | 8 | 8 | 8 | 8 | 7 | 7
Completed | 8 | 8 | 8 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Period: Third Intervention (Period 3)
Arm/Group | Group 1, Seq 1: LY2216684, Albuterol, LY2216684+Albuterol | Group 1, Seq 2: Albuterol, LY2216684+Albuterol, LY2216684 | Group 1, Seq 3: LY2216684+Albuterol, LY2216684, Albuterol | Group 2, Seq 1: LY2216684, Propranolol, LY2216684+Propranolol | Group 2, Seq 2: Propranolol, LY2216684+Propranolol, LY2216684 | Group 2, Seq 3: LY2216684+Propranolol, LY2216684, Propranolol
Started | 8 | 8 | 8 | 7 | 7 | 6
Completed | 8 | 7 | 8 | 7 | 7 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Group 1, Any Sequence (LY2216684, Albuterol, or Placebo): Participants were administered LY2216684, albuterol, or placebo during Periods 1, 2, and 3.
  LY2216684 or placebo was administered as an 18-milligram (mg) oral dose (two 9-mg tablets) once daily (QD) on Days 1 through 5 of each period.
  Albuterol or placebo was co-administered as a 2-mg oral dose (one 2-mg tablet) QD on Days 1, 3, and 5 of each period.
- Group 2, Any Sequence (LY2216684, Propranolol, or Placebo): Participants were administered LY2216684, propranolol, or placebo during Periods 1, 2, and 3.
  LY2216684 or placebo was administered as an 18-milligram (mg) oral dose (two 9-mg tablets) QD on Days 1 through 5 of each period.
  Propranolol or placebo was co-administered as a 40-mg oral dose (one 40-mg tablet) QD on Days 1, 3, and 5 of each period.
- Total: Total of all reporting groups
Arm/Group | Group 1, Any Sequence (LY2216684, Albuterol, or Placebo) | Group 2, Any Sequence (LY2216684, Propranolol, or Placebo) | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (12.0) | 36.3 (10.9) | 35.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 22 | 23 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 6 | 10 | 16
  White | 16 | 14 | 30
  More than 1 race | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 26.10 (3.40) | 28.04 (3.33) | 27.07 (3.47)

OUTCOME MEASURES:

1. Primary Outcome: Maximum, Minimum and Average Changes in Heart Rate
Description: Using a Holter monitor, heart rate was recorded every 10 minutes through 24 hours postdose on Days 1, 3, and 5 of each period. Baseline heart rate was the average of 10-minute readings taken over 2 hours prior to dosing on Day 1 of each period. Postdose heart rate was summarized over 1-hour increments using the average of the 10-minute readings within these intervals. The postdose heart rate for a day was the average heart rate for 24 hours. The least squares (LS) mean change from baseline heart rate is reported. LS mean was calculated using a mixed effects model and adjusted for participant, sequence, period, time, treatment, and time by treatment interaction.
Time Frame: Period 1, 2, 3: Baseline, Days 1 and 3 and 5 (postdose every 10 minutes through 24 hours postdose)
Population: Randomized participants with at least 1 postdose heart rate measurement.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Groups:
- LY2216684 (Group 1): Participants randomized to Group 1 who received LY2216684 administered as an 18-milligram (mg) oral dose (two 9-mg tablets) once daily (QD) on Days 1 through 5 with single oral doses of placebo (for albuterol) co-administered on Days 1, 3, and 5 in any treatment period.
- Albuterol: Participants randomized to Group 1 who received oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5 in any treatment period.
- LY2216684+Albuterol: Participants randomized to Group 1 who received LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5 in any treatment period.
- LY2216684 (Group 2): Participants randomized to Group 2 who received LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of placebo (for propranolol) co-administered on Days 1, 3, and 5 in any treatment period.
- Propranolol: Participants randomized to Group 2 who received oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 40 mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5 in any treatment period.
- LY2216684+Propranolol: Participants randomized to Group 2 who received LY2216684 administered as an 18-mg oral dose (two 9-mg tablets) QD on Days 1 through 5 with single oral doses of 40 mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5 in any treatment period.
Arm/Group | LY2216684 (Group 1) | Albuterol | LY2216684+Albuterol | LY2216684 (Group 2) | Propranolol | LY2216684+Propranolol
Number analyzed (Participants) | 24 | 24 | 24 | 22 | 22 | 22
beats per minute (bpm)
  Day 1 Maximum Change | 33.4 [29.6 to 37.2] | 15.7 [11.9 to 19.5] | 35.7 [31.9 to 39.5] | 31.1 [28.1 to 34.1] | 9.41 [6.40 to 12.4] | 17.2 [14.2 to 20.2]
  Day 1 Minimum Change | -9.23 [-11.4 to -7.05] | -15.2 [-17.4 to -13.0] | -9.03 [-11.2 to -6.86] | -5.81 [-7.97 to -3.65] | -14.8 [-17.0 to -12.6] | -10.4 [-12.6 to -8.27]
  Day 1 Average Change | 9.33 [7.08 to 11.6] | -0.788 [-3.03 to 1.46] | 10.9 [8.64 to 13.1] | 9.55 [7.50 to 11.6] | -3.94 [-6.00 to -1.89] | 1.11 [-0.934 to 3.16]
  Day 3 Maximum Change | 36.3 [32.1 to 40.4] | 19.7 [15.6 to 23.7] | 37.2 [33.0 to 41.3] | 37.2 [34.0 to 40.5] | 15.2 [12.0 to 18.4] | 27.3 [24.1 to 30.5]
  Day 3 Minimum Change | -7.05 [-9.95 to -4.15] | -16.3 [-19.1 to -13.4] | -9.76 [-12.7 to -6.86] | -5.94 [-8.45 to -3.42] | -16.1 [-18.6 to -13.6] | -9.40 [-11.9 to -6.89]
  Day 3 Average Change | 12.6 [9.82 to 15.5] | 0.102 [-2.66 to 2.87] | 14.3 [11.5 to 17.1] | 14.2 [11.9 to 16.5] | -4.34 [-6.65 to -2.03] | 6.01 [3.71 to 8.31]
  Day 5 Maximum Change | 40.4 [35.8 to 45.0] | 19.9 [15.5 to 24.3] | 39.3 [34.9 to 43.8] | 36.9 [33.5 to 40.3] | 14.0 [10.6 to 17.4] | 26.3 [22.9 to 29.7]
  Day 5 Minimum Change | -9.47 [-12.1 to -6.81] | -16.3 [-18.9 to -13.8] | -7.27 [-9.88 to -4.66] | -5.21 [-8.19 to -2.23] | -15.4 [-18.4 to -12.4] | -9.46 [-12.4 to -6.48]
  Day 5 Average Change | 14.6 [11.6 to 17.5] | 1.05 [-1.79 to 3.89] | 15.7 [12.8 to 18.6] | 15.0 [12.4 to 17.6] | -3.65 [-6.27 to -1.03] | 6.25 [3.64 to 8.86]
Statistical Analysis 1: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 2.27, 95% CI 2-sided [-3.96 to 8.49]
Statistical Analysis 2: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 0.198, 95% CI 2-sided [-3.19 to 3.59]
Statistical Analysis 3: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 1.55, 95% CI 2-sided [-2.25 to 5.35]
Statistical Analysis 4: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 20.0, 95% CI 2-sided [13.7 to 26.2]
Statistical Analysis 5: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 6.19, 95% CI 2-sided [2.80 to 9.58]
Statistical Analysis 6: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 11.7, 95% CI 2-sided [7.87 to 15.5]
Statistical Analysis 7: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -13.9, 95% CI 2-sided [-18.9 to -8.80]
Statistical Analysis 8: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -4.62, 95% CI 2-sided [-7.67 to -1.56]
Statistical Analysis 9: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -8.43, 95% CI 2-sided [-11.5 to -5.33]
Statistical Analysis 10: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 7.80, 95% CI 2-sided [2.72 to 12.9]
Statistical Analysis 11: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 4.38, 95% CI 2-sided [1.30 to 7.46]
Statistical Analysis 12: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 5.06, 95% CI 2-sided [1.93 to 8.18]
Statistical Analysis 13: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 3 where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 0.905, 95% CI 2-sided [-5.49 to 7.30]
Statistical Analysis 14: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 3 where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -2.71, 95% CI 2-sided [-6.96 to 1.54]
Statistical Analysis 15: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 1.66, 95% CI 2-sided [-2.85 to 6.16]
Statistical Analysis 16: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 3 where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 17.5, 95% CI 2-sided [11.2 to 23.8]
Statistical Analysis 17: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 6.51, 95% CI 2-sided [2.32 to 10.7]
Statistical Analysis 18: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 14.2, 95% CI 2-sided [9.75 to 18.7]
Statistical Analysis 19: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -9.98, 95% CI 2-sided [-14.6 to -5.34]
Statistical Analysis 20: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -3.46, 95% CI 2-sided [-7.22 to 0.297]
Statistical Analysis 21: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -8.16, 95% CI 2-sided [-11.6 to -4.71]
Statistical Analysis 22: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 12.1, 95% CI 2-sided [7.39 to 16.8]
Statistical Analysis 23: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 6.70, 95% CI 2-sided [2.91 to 10.5]
Statistical Analysis 24: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 10.3, 95% CI 2-sided [6.88 to 13.8]
Statistical Analysis 25: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -1.06, 95% CI 2-sided [-7.41 to 5.30]
Statistical Analysis 26: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 2.20, 95% CI 2-sided [-2.15 to 6.56]
Statistical Analysis 27: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 1.12, 95% CI 2-sided [-3.23 to 5.47]
Statistical Analysis 28: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 5 where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 19.4, 95% CI 2-sided [13.2 to 25.6]
Statistical Analysis 29: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 5 where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 9.04, 95% CI 2-sided [4.78 to 13.3]
Statistical Analysis 30: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 14.7, 95% CI 2-sided [10.4 to 18.9]
Statistical Analysis 31: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -10.6, 95% CI 2-sided [-15.6 to -5.52]
Statistical Analysis 32: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -4.25, 95% CI 2-sided [-9.26 to 0.764]
Statistical Analysis 33: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -8.76, 95% CI 2-sided [-12.6 to -4.87]
Statistical Analysis 34: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in heart rate on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 12.3, 95% CI 2-sided [7.17 to 17.4]
Statistical Analysis 35: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in heart rate on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 5.95, 95% CI 2-sided [0.917 to 11.0]
Statistical Analysis 36: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in heart rate on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 9.90, 95% CI 2-sided [5.98 to 13.8]

2. Secondary Outcome: Maximum, Minimum and Average Changes in Systolic Blood Pressure
Description: Systolic blood pressure was measured using ambulatory blood pressure monitoring (ABPM) recorded every 15 minutes during the daytime (0600 through 2200 hours) and every hour throughout the night time (2200 through 0600 hours) on Days 1, 3, and 5 of each period. Baseline systolic blood pressure was the average of 15-minute readings taken over 2 hours prior to dosing on Day 1 of each period. Postdose systolic blood pressure from ABPM was summarized over 1-hour increments using the average of the 15-minute readings within these intervals. The postdose systolic blood pressure for a day was the average systolic blood pressure for 24 hours. The least squares (LS) mean change from baseline systolic blood pressure is reported. LS mean was calculated using a mixed effects model and adjusted for participant, sequence, period, time, treatment, and time by treatment interaction.
Time Frame: Period 1, 2, 3: Baseline, Days 1 and 3 and 5 (postdose every 15 minutes from 0600 hours through 2200 hours and every hour from 2200 hours through 0600 hours)
Population: Randomized participants with at least 1 postdose systolic blood pressure measurement.
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeters of mercury (mm Hg)
Arm/Group | LY2216684 (Group 1) | Albuterol | LY2216684+Albuterol | LY2216684 (Group 2) | Propranolol | LY2216684+Propranolol
Number analyzed (Participants) | 24 | 23 | 24 | 22 | 22 | 22
millimeters of mercury (mm Hg)
  Day 1 Maximum Change | 14.1 [11.9 to 16.4] | 15.2 [12.9 to 17.5] | 15.8 [13.5 to 18.0] | 17.3 [14.3 to 20.3] | 9.39 [6.39 to 12.4] | 10.9 [7.87 to 13.8]
  Day 1 Minimum Change | -18.0 [-20.8 to -15.2] | -20.5 [-23.4 to -17.7] | -15.3 [-18.1 to -12.5] | -17.7 [-21.3 to -14.2] | -29.0 [-32.5 to -25.4] | -17.5 [-21.1 to -14.0]
  Day 1 Average Change | -0.986 [-2.97 to 0.995] | -0.912 [-2.93 to 1.11] | 1.69 [-0.292 to 3.67] | 1.73 [-0.508 to 3.97] | -8.50 [-10.7 to -6.25] | -1.35 [-3.59 to 0.884]
  Day 3 Maximum Change | 13.5 [9.99 to 16.9] | 15.6 [12.1 to 19.1] | 13.5 [10.1 to 16.9] | 15.3 [12.1 to 18.6] | 7.99 [4.74 to 11.2] | 11.2 [7.89 to 14.5]
  Day 3 Minimum Change | -19.4 [-22.3 to -16.5] | -24.9 [-27.8 to -22.0] | -20.6 [-23.4 to -17.7] | -18.5 [-21.7 to -15.3] | -27.2 [-30.4 to -24.0] | -23.3 [-26.5 to -20.0]
  Day 3 Average Change | -1.65 [-4.07 to 0.762] | -1.87 [-4.29 to 0.548] | -1.99 [-4.35 to 0.375] | 0.289 [-2.35 to 2.93] | -8.75 [-11.4 to -6.10] | -3.91 [-6.60 to -1.21]
  Day 5 Maximum Change | 13.9 [10.4 to 17.3] | 15.9 [12.5 to 19.4] | 16.2 [12.9 to 19.6] | 14.7 [11.3 to 18.0] | 11.1 [7.72 to 14.5] | 13.1 [9.69 to 16.4]
  Day 5 Minimum Change | -20.8 [-24.0 to -17.6] | -22.1 [-25.3 to -18.9] | -18.9 [-22.0 to -15.8] | -21.1 [-24.5 to -17.6] | -24.9 [-28.3 to -21.5] | -21.2 [-24.6 to -17.8]
  Day 5 Average Change | -2.07 [-4.40 to 0.270] | -2.36 [-4.69 to -0.0204] | -0.233 [-2.52 to 2.05] | -1.72 [-4.30 to 0.865] | -6.83 [-9.42 to -4.24] | -2.55 [-5.13 to 0.0363]
Statistical Analysis 1: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 1.62, 95% CI 2-sided [-1.81 to 5.06]
Statistical Analysis 2: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 2.73, 95% CI 2-sided [-1.38 to 6.85]
Statistical Analysis 3: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 2.67, 95% CI 2-sided [-0.209 to 5.56]
Statistical Analysis 4: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 0.541, 95% CI 2-sided [-2.94 to 4.02]
Statistical Analysis 5: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 5.26, 95% CI 2-sided [1.09 to 9.43]
Statistical Analysis 6: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 2.60, 95% CI 2-sided [-0.322 to 5.52]
Statistical Analysis 7: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -6.46, 95% CI 2-sided [-11.5 to -1.41]
Statistical Analysis 8: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = 0.171, 95% CI 2-sided [-5.21 to 5.56]
Statistical Analysis 9: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -3.09, 95% CI 2-sided [-6.73 to 0.557]
Statistical Analysis 10: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 1.46, 95% CI 2-sided [-3.61 to 6.53]
Statistical Analysis 11: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 11.4, 95% CI 2-sided [5.99 to 16.8]
Statistical Analysis 12: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 7.15, 95% CI 2-sided [3.49 to 10.8]
Statistical Analysis 13: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 0.0309, 95% CI 2-sided [-5.28 to 5.34]
Statistical Analysis 14: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -1.17, 95% CI 2-sided [-5.93 to 3.59]
Statistical Analysis 15: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -0.333, 95% CI 2-sided [-4.35 to 3.68]
Statistical Analysis 16: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = -2.11, 95% CI 2-sided [-7.42 to 3.20]
Statistical Analysis 17: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 4.36, 95% CI 2-sided [-0.404 to 9.12]
Statistical Analysis 18: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = -0.119, 95% CI 2-sided [-4.14 to 3.90]
Statistical Analysis 19: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -4.16, 95% CI 2-sided [-9.69 to 1.37]
Statistical Analysis 20: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -4.76, 95% CI 2-sided [-10.2 to 0.718]
Statistical Analysis 21: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -4.20, 95% CI 2-sided [-8.71 to 0.320]
Statistical Analysis 22: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 3.20, 95% CI 2-sided [-2.34 to 8.74]
Statistical Analysis 23: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 3.95, 95% CI 2-sided [-1.54 to 9.43]
Statistical Analysis 24: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 4.84, 95% CI 2-sided [0.319 to 9.37]
Statistical Analysis 25: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 2.34, 95% CI 2-sided [-3.44 to 8.12]
Statistical Analysis 26: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 1.89, 95% CI 2-sided [-3.22 to 7.00]
Statistical Analysis 27: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 1.83, 95% CI 2-sided [-1.85 to 5.52]
Statistical Analysis 28: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 0.327, 95% CI 2-sided [-5.45 to 6.10]
Statistical Analysis 29: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 3.18, 95% CI 2-sided [-1.93 to 8.29]
Statistical Analysis 30: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 2.12, 95% CI 2-sided [-1.56 to 5.81]
Statistical Analysis 31: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -1.60, 95% CI 2-sided [-6.79 to 3.59]
Statistical Analysis 32: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -0.163, 95% CI 2-sided [-5.00 to 4.68]
Statistical Analysis 33: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -0.829, 95% CI 2-sided [-5.20 to 3.54]
Statistical Analysis 34: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in systolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 1.95, 95% CI 2-sided [-3.27 to 7.17]
Statistical Analysis 35: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in systolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 3.71, 95% CI 2-sided [-1.17 to 8.59]
Statistical Analysis 36: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in systolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 4.28, 95% CI 2-sided [-0.103 to 8.67]

3. Secondary Outcome: Maximum, Minimum and Average Changes in Diastolic Blood Pressure
Description: Diastolic blood pressure was measured using ambulatory blood pressure monitoring (ABPM) recorded every 15 minutes during the daytime (0600 through 2200 hours) and every hour throughout the night time (2200 through 0600 hours) on Days 1, 3, and 5 of each period. Baseline diastolic blood pressure was the average of 15-minute readings taken over 2 hours prior to dosing on Day 1 of each period. Postdose diastolic blood pressure from ABPM was summarized over 1-hour increments using the average of the 15-minute readings within these intervals. The postdose diastolic blood pressure for a day was the average diastolic blood pressure for 24 hours. The least squares (LS) mean change from baseline diastolic blood pressure is reported. LS mean was calculated using a mixed effects model and adjusted for participant, sequence, period, time, treatment, and time by treatment interaction.
Time Frame: as for outcome 2
Population: Randomized participants with at least 1 postdose diastolic blood pressure measurement.
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeters of mercury (mm Hg)
Arm/Group | LY2216684 (Group 1) | Albuterol | LY2216684+Albuterol | LY2216684 (Group 2) | Propranolol | LY2216684+Propranolol
Number analyzed (Participants) | 24 | 23 | 24 | 22 | 22 | 22
millimeters of mercury (mm Hg)
  Day 1 Maximum Change | 13.4 [11.7 to 15.2] | 10.8 [9.05 to 12.6] | 12.2 [10.5 to 13.9] | 14.9 [12.6 to 17.1] | 8.16 [5.88 to 10.4] | 10.6 [8.37 to 12.9]
  Day 1 Minimum Change | -17.3 [-19.4 to -15.1] | -19.9 [-22.1 to -17.7] | -16.2 [-18.4 to -14.1] | -17.9 [-21.2 to -14.6] | -26.7 [-30.0 to -23.4] | -17.6 [-20.9 to -14.3]
  Day 1 Average Change | -0.674 [-2.38 to 1.03] | -3.27 [-5.01 to -1.53] | -0.873 [-2.58 to 0.833] | 0.481 [-1.37 to 2.33] | -7.47 [-9.33 to -5.61] | -1.44 [-3.29 to 0.410]
  Day 3 Maximum Change | 13.6 [11.4 to 15.9] | 11.8 [9.60 to 14.1] | 12.7 [10.5 to 14.9] | 15.4 [13.0 to 17.7] | 6.87 [4.51 to 9.24] | 12.5 [10.1 to 14.9]
  Day 3 Minimum Change | -18.1 [-21.0 to -15.3] | -21.5 [-24.3 to -18.7] | -18.6 [-21.4 to -15.8] | -17.8 [-20.5 to -15.2] | -26.6 [-29.3 to -24.0] | -18.8 [-21.5 to -16.1]
  Day 3 Average Change | -0.537 [-2.24 to 1.17] | -3.10 [-4.80 to -1.40] | -0.159 [-1.83 to 1.51] | 0.619 [-1.44 to 2.68] | -7.80 [-9.87 to -5.74] | -1.20 [-3.31 to 0.900]
  Day 5 Maximum Change | 13.8 [11.3 to 16.4] | 12.8 [10.2 to 15.3] | 14.7 [12.2 to 17.2] | 13.1 [10.2 to 16.0] | 6.58 [3.69 to 9.47] | 13.8 [11.0 to 16.7]
  Day 5 Minimum Change | -17.0 [-20.2 to -13.8] | -21.6 [-24.8 to -18.4] | -20.5 [-23.7 to -17.3] | -19.1 [-22.2 to -15.9] | -26.6 [-29.7 to -23.4] | -21.0 [-24.2 to -17.8]
  Day 5 Average | 0.233 [-1.74 to 2.20] | -3.17 [-5.14 to -1.20] | -0.140 [-2.08 to 1.80] | -0.631 [-2.81 to 1.55] | -7.33 [-9.52 to -5.14] | -1.80 [-3.99 to 0.381]
Statistical Analysis 1: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -1.23, 95% CI 2-sided [-3.90 to 1.44]
Statistical Analysis 2: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 1.05, 95% CI 2-sided [-1.91 to 4.02]
Statistical Analysis 3: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -0.199, 95% CI 2-sided [-2.58 to 2.18]
Statistical Analysis 4: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 1.37, 95% CI 2-sided [-1.34 to 4.07]
Statistical Analysis 5: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 3.68, 95% CI 2-sided [0.674 to 6.69]
Statistical Analysis 6: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 1, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 2.40, 95% CI 2-sided [-0.0178 to 4.81]
Statistical Analysis 7: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -4.22, 95% CI 2-sided [-7.83 to -0.619]
Statistical Analysis 8: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = 0.335, 95% CI 2-sided [-4.45 to 5.12]
Statistical Analysis 9: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -1.92, 95% CI 2-sided [-4.81 to 0.969]
Statistical Analysis 10: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 2.47, 95% CI 2-sided [-1.15 to 6.10]
Statistical Analysis 11: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 9.12, 95% CI 2-sided [4.30 to 13.9]
Statistical Analysis 12: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 1, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 6.03, 95% CI 2-sided [3.12 to 8.94]
Statistical Analysis 13: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -0.913, 95% CI 2-sided [-4.65 to 2.82]
Statistical Analysis 14: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -0.444, 95% CI 2-sided [-4.33 to 3.44]
Statistical Analysis 15: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 0.378, 95% CI 2-sided [-2.20 to 2.95]
Statistical Analysis 16: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 0.878, 95% CI 2-sided [-2.86 to 4.62]
Statistical Analysis 17: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 2.92, 95% CI 2-sided [-0.966 to 6.80]
Statistical Analysis 18: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 3, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 2.94, 95% CI 2-sided [0.366 to 5.52]
Statistical Analysis 19: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -2.88, 95% CI 2-sided [-6.84 to 1.07]
Statistical Analysis 20: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -0.975, 95% CI 2-sided [-5.39 to 3.44]
Statistical Analysis 21: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -1.82, 95% CI 2-sided [-5.30 to 1.66]
Statistical Analysis 22: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 5.60, 95% CI 2-sided [1.63 to 9.56]
Statistical Analysis 23: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 7.82, 95% CI 2-sided [3.39 to 12.3]
Statistical Analysis 24: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 3, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 6.60, 95% CI 2-sided [3.11 to 10.1]
Statistical Analysis 25: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = 0.847, 95% CI 2-sided [-3.23 to 4.92]
Statistical Analysis 26: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -3.48, 95% CI 2-sided [-8.17 to 1.21]
Statistical Analysis 27: Comparison: LY2216684 (Group 1) vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the LY2216684 (Group 1) treatment arm; Test type: Superiority or Other; LS mean difference = -0.372, 95% CI 2-sided [-2.88 to 2.14]
Statistical Analysis 28: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 1.90, 95% CI 2-sided [-2.17 to 5.98]
Statistical Analysis 29: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 1.07, 95% CI 2-sided [-3.62 to 5.76]
Statistical Analysis 30: Comparison: Albuterol vs LY2216684+Albuterol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 5, where test is the LY2216684+albuterol treatment arm and reference is the albuterol treatment arm; Test type: Superiority or Other; LS mean difference = 3.03, 95% CI 2-sided [0.522 to 5.55]
Statistical Analysis 31: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = 0.737, 95% CI 2-sided [-3.90 to 5.38]
Statistical Analysis 32: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -1.95, 95% CI 2-sided [-6.36 to 2.47]
Statistical Analysis 33: Comparison: LY2216684 (Group 2) vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the LY2216684 (Group 2) treatment arm; Test type: Superiority or Other; LS mean difference = -1.17, 95% CI 2-sided [-4.79 to 2.45]
Statistical Analysis 34: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the maximum changes in diastolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 7.25, 95% CI 2-sided [2.59 to 11.9]
Statistical Analysis 35: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the minimum changes in diastolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 5.58, 95% CI 2-sided [1.13 to 10.0]
Statistical Analysis 36: Comparison: Propranolol vs LY2216684+Propranolol; Difference of LS means (test minus reference) for the average changes in diastolic blood pressure on Day 5, where test is the LY2216684+propranolol treatment arm and reference is the propranolol treatment arm; Test type: Superiority or Other; LS mean difference = 5.53, 95% CI 2-sided [1.89 to 9.16]

ADVERSE EVENTS:
Groups:
- Albuterol: Participants randomized to Group 1 who received who received oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 2 mg albuterol (one 2-mg tablet) co-administered on Days 1, 3, and 5 in any treatment period.
- Propranolol: Participants randomized to Group 2 who received oral doses of placebo (for LY2216684) administered QD on Days 1 through 5 with single oral doses of 40-mg propranolol (one 40-mg tablet) co-administered on Days 1, 3, and 5 in any treatment period.
Arm/Group | LY2216684 (Group 1) | Albuterol | LY2216684+Albuterol | LY2216684 (Group 2) | Propranolol | LY2216684+Propranolol
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 13/24 | 2/24 | 13/24 | 9/22 | 8/22 | 13/22
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 (Group 1) (N=24) | Albuterol (N=24) | LY2216684+Albuterol (N=24) | LY2216684 (Group 2) (N=22) | Propranolol (N=22) | LY2216684+Propranolol (N=22)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (2) | 4 (4) | 0 (0) | 3 (3) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/7 (0) | 0/7 (0) | 0/7 (0) | 0/10 (0) | 1/10 (1) | 0/9 (0)
Genital pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 0/17 (0) | 0/17 (0) | 0/17 (0) | 1/12 (1) | 0/12 (0) | 0/13 (0)
Penile size reduced (Reproductive system and breast disorders) | 0/17 (0) | 0/17 (0) | 1/17 (1) | 0/12 (0) | 0/12 (0) | 1/13 (1)
Scrotal pain (Reproductive system and breast disorders) | 1/17 (1) | 0/17 (0) | 0/17 (0) | 0/12 (0) | 0/12 (0) | 0/13 (0)
Testicular pain (Reproductive system and breast disorders) | 0/17 (0) | 0/17 (0) | 0/17 (0) | 1/12 (1) | 0/12 (0) | 0/13 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days